CLINICAL TRIAL: NCT01302847
Title: Phase I/II, Multi-Center, Open-Label Pharmacokinetic, Safety, Tolerability and Antiviral Activity of Dolutegravir, a Novel Integrase Inhibitor, in Combination Regimens in HIV-1 Infected Infants, Children and Adolescents
Brief Title: Safety of and Immune Response to Dolutegravir in HIV-1 Infected Infants, Children, and Adolescents
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P1093; 11773 (Registry Identifier: DAIDS-ES); 2010-020988-20 (EudraCT Number); IMPAACT P1093
Record Dates: First submitted 2011-02-15; First posted 2011-02-24 (Estimated); Results first posted 2022-03-22 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-10

CONDITIONS: HIV Infections
Keywords: Integrase Inhibitors; Infant; Child; Adolescent
MeSH Terms: conditions — HIV Infections | interventions — Suspensions; dolutegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Cohort I (Experimental): Adolescents 12 to younger than 18 years of age who received DTG film-coated tablets
  Interventions: Drug: DTG film-coated tablets
- Cohort IIA (Experimental): Children 6 to younger than 12 years of age who received DTG film-coated tablets
  Interventions: Drug: DTG film-coated tablets
- Cohort IIB (Experimental): Children 6 to younger than 12 years of age who received DTG granules for suspension
  Interventions: Drug: DTG granules for suspension
- Cohort III (Experimental): Children 2 to younger than 6 years of age who received DTG granules for suspension
  Interventions: Drug: DTG granules for suspension
- Cohort IV (Experimental): Children 6 months to younger than 2 years of age who received DTG granules for suspension
  Interventions: Drug: DTG granules for suspension
- Cohort III-DT (Experimental): Children 2 to younger than 6 years of age who received DTG dispersible tablets
  Interventions: Drug: DTG dispersible tablets
- Cohort IV-DT (Experimental): Children 6 months to younger than 2 years of age who received DTG dispersible tablets
  Interventions: Drug: DTG dispersible tablets
- Cohort V-DT (Experimental): Infants 4 weeks to younger than 6 months of age who received DTG dispersible tablets
  Interventions: Drug: DTG dispersible tablets

INTERVENTIONS:
Drug: DTG film-coated tablets — DTG film-coated tablets initial starting dose at ~1 mg/kg with a maximum dose of 50 mg; orally once daily. Participants weighing ≥ 35kg received the proposed dose of 50 mg of DTG film-coated tablets.
  Arms: Cohort I; Cohort IIA
Drug: DTG granules for suspension — DTG granules for suspension initial starting dose at ~0.64 mg/kg with a maximum dose of 32 mg; orally once daily.
  Arms: Cohort IIB; Cohort III; Cohort IV
Drug: DTG dispersible tablets — DTG dispersible tablets initial starting dose of ~0.8 mg/kg with a maximum dose of 30 mg; orally once daily. The proposed weight-band dosing was:
  Weight band 3 to <6 kg: 5 mg DTG dispersible tablets; Weight band 6 to <10 kg: 15 mg DTG dispersible tablets; Weight band 10 to <14 kg: 20 mg DTG dispersible tablets; Weight band 14 to <20 kg: 25 mg DTG dispersible tablets; Weight band ≥20 kg: 30 mg DTG dispersible tablets.
  Arms: Cohort III-DT
Drug: DTG dispersible tablets — DTG dispersible tablets initial starting dose of ~1.25 mg/kg with a maximum dose of 30 mg; orally once daily. The proposed weight-band dosing was:
  Weight band 3 to <6 kg: 5 mg DTG dispersible tablets; Weight band 6 to <10 kg: 15 mg DTG dispersible tablets; Weight band 10 to <14 kg: 20 mg DTG dispersible tablets; Weight band 14 to <20 kg: 25 mg DTG dispersible tablets; Weight band ≥20 kg: 30 mg DTG dispersible tablets.
  Arms: Cohort IV-DT
Drug: DTG dispersible tablets — DTG dispersible tablets initial starting dose of ~1.25 mg/kg with a maximum dose of 30 mg; orally once daily. The proposed weight-band dosing was:
  Weight band 3 to <6 kg: 5 mg DTG dispersible tablets; Weight band 6 to <10 kg: 15 mg DTG dispersible tablets.
  Arms: Cohort V-DT

SUMMARY:
Dolutegravir (DTG) is an HIV drug in the integrase inhibitor drug class. This study evaluated the pharmacokinetics (PK), safety, tolerability of and immune response to DTG when used concurrently with optimized background therapy (OBT) in HIV-1 infected infants, children, and adolescents.

DETAILED DESCRIPTION:
DTG is an HIV medicine in the integrase inhibitor drug class. The purpose of this study was to evaluate the pharmacokinetics, safety, tolerability, and antiviral activity of DTG when used concurrently with OBT in HIV-1 infected infants, children, and adolescents.

Participants in this study were evaluated for PK, safety and tolerability through 48 weeks, followed by additional long-term study follow-up that lasted for approximately 144 weeks (3 years), for a total of 192 weeks on study. This study had two stages. Stage I provided pharmacokinetics, short-term tolerability and safety data on DTG on a limited number of participants to permit dose selection for further study in Stage II. Once a Stage I dose was accepted, enrollment to Stage II began to complete enrollment to the cohort. Stage II provided longer-term safety and antiviral activity data among a larger number of participants.

Infants, children and adolescents with HIV-1, aged ≥ 4 weeks to < 18 years enrolled in the age and formulation cohorts specified below:

* Cohort I: Adolescents ≥ 12 to <18 years of age (film-coated tablets)
* Cohort IIA: Children ≥ 6 to <12 years of age (film-coated tablets)
* Cohort IIB: Children ≥ 6 to <12 years of age (granules for suspension)
* Cohort III: Children ≥ 2 to < 6 years of age (granules for suspension)
* Cohort IV: Children ≥ 6 months to < 2 years of age (granules for suspension)
* Cohort III-DT: Children ≥ 2 to < 6 years of age (dispersible tablets)
* Cohort IV-DT: Children ≥ 6 months to < 2 years of age (dispersible tablets)
* Cohort V-DT: Infants ≥ 4 weeks to < 6 months (dispersible tablets)

Cohorts were opened sequentially according by age group (starting with the older age group), DTG formulation, and study stage, i.e. Initial study enrollment was for Cohort I and progressed to Cohort IIA once Cohort I Stage I met the PK and safety criteria, followed by opening of Cohort IIB. Each cohort enrolled in two sequential stages: Stage I and II (the only exception is Cohort IIB, which only enrolled through Stage I). Sequential enrollment for Cohort III and IV proceeded in the same manner. Cohort V never enrolled because of the recommended changes in dosing and inclusion of enrollment weight band in the criteria for dose finding.

Stage I participants had physical examinations and had blood draws for safety assessments at study visits: Day 0; Day 5 (+5 days); and Weeks 4, 8, 12, 16, 24, 32, 40, and 48. Stage I participants also had intensive PK sampling with blood samples collected at time 0 (pre-dose), and at 1, 2, 3, 4, 6, 8 and 24 hours post dosing. Once a Stage I treatment dose was accepted, enrollment to Stage II began to complete enrollment to the cohort. Stage II participants had physical examinations and blood draws for safety assessment at study visits: Day 0; Day 10; and Weeks 4, 8, 12, 16, 24, 32, 40, and 48. Blood, plasma, and urine were collected and tested to measure immune response. Females of childbearing potential underwent pregnancy testing at screening and at every study visit.

After 48 weeks, all Stage I and Stage II participants entered the long-term study follow-up and continued to receive DTG. During this time, participants had safety and/or antiviral activity assessments every 12 weeks for up to 3 years.

The study was able to determine a proposed dose (i.e. optimal dose) for Cohorts I, IIA, III-DT, IV-DT, and V-DT but not for Cohorts IIB, III, and IV. Participants on the proposed dose had intensive PK sampling between days 5 and10 of DTG initiation with blood samples collected at time 0 (pre-dose), and at 1, 2, 3, 4, 6, 8 and 24 hours post dosing.

The study is closed to accrual and study follow-up was completed on Oct 18, 2023.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HIV-1 infection, defined as positive results from two samples collected at different time points (see protocol for more information)
* Participant belonged to one of the ARV exposure groups below:

  1. ARV-treatment experienced (not including receipt of ARVs as prophylaxis or for prevention of perinatal transmission)

     * Previously took ARVs for treatment, but not taking ARVs at study screening.
     * Had been off treatment for greater than or equal to 4 weeks prior to screening, OR
     * At screening, taking ARVs for treatment but failing.
     * Was on an unchanged, failing therapeutic regimen within the 4 to 12 weeks prior to screening (less than or equal to 1 log drop in HIV-1 RNA within the 4 to 12 weeks prior to screening). OR
     * For participants less than 2 years of age, initiated ARVs for treatment less than 4 weeks prior to screening.
  2. ARV treatment naive (no exposure to ARVs for treatment; could have received ARVs for prophylaxis or prevention of perinatal transmission)
* If an infant had received nevirapine (NVP) as prophylaxis to prevent perinatal transmission, he or she did not receive NVP for at least 14 days prior to enrollment into Stage I or II.
* HIV-1 RNA viral load greater than 1,000 copies/mL of plasma at screening.
* Demonstrated ability or willingness to swallow assigned study medications.
* Parent or legal guardian were able and willing to provide signed informed consent.
* Female participants of reproductive potential, defined as having reached menarche, and who were engaging in sexual activity that could lead to pregnancy, agreed to use two contraceptive methods while on study and for two weeks after stopping study drug.
* Males engaging in sexual activity that could lead to HIV-1 transmission agreed to use a condom.
* Agreed to stay on optimized background therapy (OBT) while on study:

  * Participants who at screening were greater than or equal to 2 years of age and ARV-treatment experienced, had at screening at least one fully active drug for the OBT.
  * Participants who were greater than or equal to 2 years of age and ARV-treatment naïve, had genotype testing at screening/entry even with results pending.
  * Participants less than 2 years of age (either ARV-treatment experienced or ARV treatment naïve), had genotype testing at screening/entry even with results pending.

Exclusion Criteria:

* Presence of any active AIDS-defining opportunistic infection
* At enrollment, participant less than 3.0 kg
* Known Grade 3 or greater of any of the following laboratory toxicities within 30 days prior to study entry: neutrophil count, hemoglobin, platelets, aspartate aminotransferase (AST), alanine transaminase (ALT), lipase, serum creatinine and total bilirubin. A single repeat within the 30 days is allowed for eligibility determination. NOTE: Grade 3 total bilirubin was allowable, if the participant was on atazanavir (ATV).
* ANY known Grade 4 laboratory toxicities within 30 days prior to study entry. NOTE: Grade 4 total bilirubin was allowable, if the participant was on ATV.
* The following liver toxicities within 30 days prior to study entry: ALT greater than 3x the upper limit of normal (ULN) AND direct bilirubin was greater than 2x ULN
* Any prior history of malignancy, with the exception of localized malignancies such as squamous cell or basal cell carcinoma of the skin
* Clinical or symptomatic evidence of pancreatitis, as determined by the clinician
* Use of any disallowed medications at time of screening (see the protocol for a complete list of disallowed medications)
* Known history of exposure to integrase inhibitor treatment by the participant or participant's mother prior to delivery/cessation of breastfeeding
* Known resistance to an integrase inhibitor
* Women who were pregnant or breastfeeding
* At screening/entry, participating in or had participated in a study with a compound or device that was not commercially available within 30 days of signing informed consent, unless permission from both Protocol Teams was granted
* Participant was unlikely to adhere to the study procedures, keep appointments, or was planning to relocate during the study to a non-IMPAACT study site
* Any clinically significant diseases (other than HIV infection) or clinically significant findings during the screening medical history or physical examination that, in the investigator's opinion, would compromise the outcome of this study
* At screening/entry had used, or anticipated using, chronic systemic immunosuppressive agents or systemic interferon (e.g., for treatment of hepatitis C virus [HCV] infection) within 30 days prior to beginning DTG study treatment. Systemic corticosteroids (e.g., prednisone or equivalent up to 2 mg/kg/day) for replacement therapy or short courses (less than or equal to 30 days) were permitted. (See protocol for more information on disallowed medications.)
* Any condition that in the opinion of the site investigator, placed the participant at an unacceptable risk of injury or render the participant unable to meet the requirements of the protocol.
* Active tuberculosis (TB) disease and/or requirement for treatment that included rifampin at the time of the screening visit. However, participants who needed rifampin treatment while on DTG were allowed to continue in P1093 provided the DTG dose was adjusted according to the protocol.

Ages: 4 Weeks to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 181 (Actual)
Dates: Start 2011-04-20 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2023-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Wiznia, M.D., Study Chair — Jacobi Medical Center; Theodore Ruel, M.D., Study Chair — University of California, San Francisco
Locations (33):
- United States (17):
  - University of California, UC San Diego CRS- Mother-Child-Adolescent HIV Program (Site ID: 4601), La Jolla, California
  - Miller Children's Hosp. Long Beach CA NICHD CRS (Site ID: 5093), Long Beach, California
  - David Geffen School of Medicine at UCLA NICHD CRS (Site ID: 5112), Los Angeles, California
  - Univ. of California San Francisco NICHD CRS (Site ID: 5091), San Francisco, California
  - Univ. of Colorado Denver NICHD CRS (Site ID: 5052), Aurora, Colorado
  - Howard Univ. Washington DC NICHD CRS (Site ID: 5044), Washington D.C., District of Columbia
  - South Florida CDTC Ft Lauderdale NICHD CRS (Site ID: 5055), Fort Lauderdale, Florida
  - USF - Tampa NICHD CRS (Site ID: 5018), Tampa, Florida
  - Rush Univ. Cook County Hosp. Chicago NICHD CRS (Site ID: 5083), Chicago, Illinois
  - Lurie Children's Hospital of Chicago (LCH) CRS (Site ID: 4001), Chicago, Illinois
  - Children's Hosp. of Boston NICHD CRS (Site ID: 5009), Boston, Massachusetts
  - Boston Medical Center Ped. HIV Program NICHD CRS (Site ID: 5011), Boston, Massachusetts
  - Metropolitan Hosp. NICHD CRS (Site ID: 5003), New York, New York
  - Bronx-Lebanon Hospital Center NICHD CRS (Site ID: 5114), The Bronx, New York
  - Jacobi Med. Ctr. Bronx NICHD CRS (Site ID: 5013), The Bronx, New York
  - DUMC Ped. CRS (Site ID: 4701), Durham, North Carolina
  - Seattle Children's Research Institute CRS (Site ID: 5017), Seattle, Washington
- Botswana (2):
  - Gaborone CRS (Site ID: 12701), Gaborone, South-East District
  - Molepolole CRS (Site ID: 12702), Gaborone
- Brazil (5):
  - SOM Federal University Minas Gerais Brazil NICHD CRS (Site ID: 5073), Belo Horizonte, Minas Gerais
  - Hospital Federal dos Servidores do Estado NICHD CRS (Site ID: 5072), Rio de Janeiro
  - Instituto de Puericultura e Pediatria Martagao Gesteira - UFRJ NICHD CRS (Site ID: 5071), Rio de Janeiro
  - Hosp. Geral De Nova Igaucu Brazil NICHD CRS (Site ID: 5097), Rio de Janeiro
  - Univ. of Sao Paulo Brazil NICHD CRS (Site ID: 5074), São Paulo
- Kenya Medical Research Institute / Walter Reed Project Clinical Research Center, Kericho CRS (Site ID: 5121), Kericho, Kenya
- South Africa (3):
  - Wits RHI Shandukani Research Centre CRS (Site ID: 8051), Johannesburg, Gauteng
  - Umlazi CRS (Site ID: 30300), Durban, KwaZulu-Natal
  - FAMCRU CRS (Site ID: 8950), Tygerberg, Western Cape
- Kilimanjaro Christian Medical Centre (KCMC) (Site ID: 5118), Moshi, Tanzania
- Thailand (3):
  - Siriraj Hospital, Mahidol University NICHD CRS (Site ID: 5115), Bangkok, Bangkoknoi
  - Chiangrai Prachanukroh Hospital NICHD CRS (Site ID: 5116), Chiang Mai
  - Chiang Mai University HIV Treatment (CMU HIV Treatment) CRS (Site ID: 31784), Chiang Mai
- Harare Family Care CRS (Site ID: 31890), Harare, Zimbabwe

REFERENCES:
- [Background] Bennetto-Hood C, Tabolt G, Savina P, Acosta EP. A sensitive HPLC-MS/MS method for the determination of dolutegravir in human plasma. J Chromatogr B Analyt Technol Biomed Life Sci. 2014 Jan 15;945-946:225-32. doi: 10.1016/j.jchromb.2013.11.054. Epub 2013 Dec 3. PMID 24361860
- [Background] Viani RM, Alvero C, Fenton T, Acosta EP, Hazra R, Townley E, Steimers D, Min S, Wiznia A; P1093 Study Team. Safety, Pharmacokinetics and Efficacy of Dolutegravir in Treatment-experienced HIV-1 Infected Adolescents: Forty-eight-week Results from IMPAACT P1093. Pediatr Infect Dis J. 2015 Nov;34(11):1207-13. doi: 10.1097/INF.0000000000000848. PMID 26244832
- [Background] Viani RM, Ruel T, Alvero C, Fenton T, Acosta EP, Hazra R, Townley E, Palumbo P, Buchanan AM, Vavro C, Singh R, Graham B, Anthony P, George K, Wiznia A; P1093 Study Team. Long-Term Safety and Efficacy of Dolutegravir in Treatment-Experienced Adolescents With Human Immunodeficiency Virus Infection: Results of the IMPAACT P1093 Study. J Pediatric Infect Dis Soc. 2020 Apr 30;9(2):159-165. doi: 10.1093/jpids/piy139. PMID 30951600
- [Derived] Ruel TD, Acosta EP, Liu JP, Gray KP, George K, Montanez N, Popson S, Buchanan AM, Bartlett M, Dayton D, Anthony P, Brothers C, Vavro C, Singh R, Koech L, Vhembo T, Mmbaga BT, Pinto JA, Dobbels EFM, Archary M, Chokephaibulkit K, Ounchanum P, Deville JG, Hazra R, Townley E, Wiznia A; IMPAACT P1093 team. Pharmacokinetics, safety, tolerability, and antiviral activity of dolutegravir dispersible tablets in infants and children with HIV-1 (IMPAACT P1093): results of an open-label, phase 1-2 trial. Lancet HIV. 2022 May;9(5):e332-e340. doi: 10.1016/S2352-3018(22)00044-3. PMID 35489377
- [Derived] Singh RP, Adkison KK, Baker M, Parasrampuria R, Wolstenholme A, Davies M, Sewell N, Brothers C, Buchanan AM. Development of Dolutegravir Single-entity and Fixed-dose Combination Formulations for Children. Pediatr Infect Dis J. 2022 Mar 1;41(3):230-237. doi: 10.1097/INF.0000000000003366. PMID 34817414
- [Derived] Vavro C, Ruel T, Wiznia A, Montanez N, Nangle K, Horton J, Buchanan AM, Stewart EL, Palumbo P. Emergence of Resistance in HIV-1 Integrase with Dolutegravir Treatment in a Pediatric Population from the IMPAACT P1093 Study. Antimicrob Agents Chemother. 2022 Jan 18;66(1):e0164521. doi: 10.1128/AAC.01645-21. Epub 2021 Oct 25. PMID 34694878
- See also: The Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 1.0, December 2004 (Clarification, August 2009). — https://rsc.niaid.nih.gov/clinical-research-sites/daids-adverse-event-grading-tables
- See also: Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual), Version 2.0, January 2010 — https://rsc.niaid.nih.gov/clinical-research-sites/manual-expedited-reporting-adverse-events-daids

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from April 20, 2011 to February 19, 2020. Participants were recruited from 9 countries in North America, South America, Africa, and Asia.
Pre-assignment Details: There was no study randomization. A participant was enrolled to a cohort based on their age at study entry.
Groups:
- Cohort I: Adolescents 12 to younger than 18 years of age who received DTG film-coated tablets.
  DTG film-coated tablets initial starting dose at ~1 mg/kg with a maximum dose of 50 mg; orally once daily.
- Cohort IIA: Children 6 to younger than 12 years of age who received DTG film-coated tablets.
  DTG film-coated tablets initial starting dose at ~1 mg/kg with a maximum dose of 50 mg; orally once daily.
- Cohort IIB: Children 6 to younger than 12 years of age who received DTG granules for suspension.
  DTG granules for suspension initial starting dose at ~0.64 mg/kg with a maximum dose of 32 mg; orally once daily.
- Cohort III: Children 2 to younger than 6 years of age who received DTG granules for suspension.
  DTG granules for suspension initial starting dose at ~0.64 mg/kg with a maximum dose of 32 mg; orally once daily.
- Cohort IV: Children 6 months to younger than 2 years of age who received DTG granules for suspension.
  DTG granules for suspension initial starting dose at ~0.64 mg/kg with a maximum dose of 32 mg; orally once daily.
- Cohort III-DT: Children 2 to younger than 6 years of age who received DTG dispersible tablets.
  DTG dispersible tablets initial starting dose of ~0.8 mg/kg with a maximum dose of 30 mg; orally once daily.
- Cohort IV-DT: Children 6 months to younger than 2 years of age who received DTG dispersible tablets.
  DTG dispersible tablets initial starting dose of ~1.25 mg/kg with a maximum dose of 30 mg; orally once daily.
- Cohort V-DT: Infants 4 weeks to younger than 6 months of age who received DTG dispersible tablets.
  DTG dispersible tablets initial starting dose of ~1.25 mg/kg with a maximum dose of 30 mg; orally once daily.
Period: Overall Study
Arm/Group | Cohort I | Cohort IIA | Cohort IIB | Cohort III | Cohort IV | Cohort III-DT | Cohort IV-DT | Cohort V-DT
Started | 23 | 23 | 15 | 17 | 7 | 36 | 35 | 25
Completed | 10 | 16 | 14 | 15 | 5 | 31 | 30 | 20
Not Completed | 13 | 7 | 1 | 2 | 2 | 5 | 5 | 5
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Pregnancy | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Virologic failure | 0 | 2 | 0 | 2 | 1 | 3 | 1 | 2
Not completed — Severe debilitation, unable to continue | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Not able to get to clinic | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Site closing | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Not willing to adhere to requirements | 5 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Not completed — Site unable to contact participant | 2 | 1 | 0 | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Participants who received at least one dose of DTG.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort I | Cohort IIA | Cohort IIB | Cohort III | Cohort IV | Cohort III-DT | Cohort IV-DT | Cohort V-DT | Total
Number analyzed (Participants) | 23 | 23 | 15 | 17 | 7 | 36 | 35 | 25 | 181
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.26 (1.79) | 8.96 (1.99) | 7.73 (1.79) | 3.59 (1.00) | 1.14 (0.41) | 3.25 (1.18) | 1.13 (0.44) | 0.03 (0.01) | 4.84 (4.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 7 | 3 | 8 | 5 | 13 | 20 | 12 | 86
  Male | 5 | 16 | 12 | 9 | 2 | 23 | 15 | 13 | 95
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 4 | 8 | 1 | 6 | 4 | 2 | 37
  Not Hispanic or Latino | 16 | 13 | 6 | 6 | 6 | 28 | 31 | 23 | 129
  Unknown or Not Reported | 1 | 4 | 5 | 3 | 0 | 2 | 0 | 0 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 3 | 3 | 2 | 3 | 7 | 1 | 3 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 12 | 12 | 10 | 11 | 3 | 25 | 30 | 20 | 123
  White | 7 | 3 | 0 | 2 | 0 | 1 | 2 | 0 | 15
  More than one race | 0 | 1 | 0 | 1 | 0 | 3 | 2 | 2 | 9
  Unknown or Not Reported | 1 | 3 | 2 | 1 | 1 | 0 | 0 | 0 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 16 | 5 | 5 | 0 | 3 | 2 | 0 | 51
  Botswana | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 5
  Tanzania | 0 | 0 | 0 | 1 | 0 | 3 | 3 | 3 | 10
  Brazil | 0 | 0 | 2 | 5 | 1 | 6 | 2 | 3 | 19
  South Africa | 0 | 4 | 6 | 4 | 2 | 6 | 4 | 2 | 28
  Uganda | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3
  Zimbabwe | 0 | 0 | 0 | 0 | 0 | 3 | 15 | 10 | 28
  Kenya | 0 | 0 | 0 | 0 | 0 | 8 | 5 | 1 | 14
  Thailand | 3 | 3 | 2 | 2 | 3 | 6 | 1 | 3 | 23
Weight [Mean (Standard Deviation); unit: kg] | 55.1 (15.6) | 30.1 (10.4) | 23.0 (4.6) | 14.4 (2.9) | 8.4 (2.0) | 13.7 (2.6) | 8.5 (1.8) | 5.7 (1.1) | 19.6 (17.0)
Height [Mean (Standard Deviation); unit: cm] | 155.4 (8.9) | 131.1 (14.0) | 121.2 (9.6) | 95.9 (8.7) | 71.0 (6.0) | 93.4 (8.9) | 71.9 (5.7) | 59.2 (3.7) | 98.9 (32.4)
CD4 Cell Count [Median (Inter-Quartile Range); unit: cells/mm^3] — Population: Participants who had non-missing values were summarized. One participant in Cohort IV had missing value.
  cells/mm^3
    number analyzed (Participants) | 23 | 23 | 15 | 17 | 6 | 36 | 35 | 25 | 180
    (all) | 466.0 [297 to 771] | 645.0 [466 to 732] | 749.0 [306 to 1041] | 900.0 [565 to 1399] | 1482.5 [1190 to 1827] | 1049.5 [559.5 to 1883] | 2121.0 [1422 to 2384] | 1916.0 [1357 to 2680] | 1053.0 [618 to 1914.5]
CD4 Percent [Median (Inter-Quartile Range); unit: Percentage of total lymphocytes] — Population: Participants who had non-missing values were summarized. One participant in Cohort IV had missing value.
  Percentage of total lymphocytes
    number analyzed (Participants) | 23 | 23 | 15 | 17 | 6 | 36 | 35 | 25 | 180
    (all) | 22.0 [18.4 to 29.2] | 24.0 [14.3 to 28.7] | 25.3 [20 to 33] | 25.0 [20 to 31] | 20.7 [14.6 to 31.1] | 24.0 [17.2 to 31.1] | 24.2 [19.8 to 32.2] | 22.7 [20.6 to 30.4] | 24.0 [18.3 to 31]
CD8 Cell Count [Median (Inter-Quartile Range); unit: cells/mm^3] — Population: Participants who had non-missing values were summarized. One participant in Cohort IV had missing value.
  cells/mm^3
    number analyzed (Participants) | 23 | 23 | 15 | 17 | 6 | 36 | 35 | 25 | 180
    (all) | 1009.0 [788 to 1303] | 1089.0 [955 to 1774] | 1103.0 [948 to 1757] | 1730.0 [1148 to 1991] | 1888.5 [1441 to 2796] | 1725.0 [1258 to 2561.5] | 2922.0 [2050 to 4546] | 2435.0 [1468 to 3789] | 1679.0 [1074.5 to 2725]
CD8 Percent [Median (Inter-Quartile Range); unit: Percentage of total lymphocytes] — Population: Participants who had non-missing values were summarized. One participant in Cohort IV had missing value.
  Percentage of total lymphocytes
    number analyzed (Participants) | 23 | 23 | 15 | 17 | 6 | 36 | 35 | 25 | 180
    (all) | 49.5 [43.8 to 59] | 53.0 [43 to 58.6] | 48.0 [44 to 51] | 39.7 [35.1 to 49.3] | 28.5 [18.2 to 34.4] | 42.2 [29.5 to 50.2] | 39.4 [31.3 to 47.2] | 31.6 [24 to 41.8] | 43.0 [32 to 50.8]
Baseline Plasma HIV-1 RNA (copies/mL) [Count of Participants; unit: Participants]
  <400 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 1 | 6
  400 - <1,000 | 0 | 1 | 0 | 0 | 1 | 3 | 1 | 0 | 6
  1,000 - <5,000 | 2 | 3 | 1 | 2 | 0 | 5 | 7 | 7 | 27
  5,000 - <10,000 | 4 | 1 | 1 | 1 | 0 | 1 | 4 | 3 | 15
  10,000 - <25,000 | 8 | 0 | 3 | 0 | 0 | 4 | 4 | 2 | 21
  25,000 - <50,000 | 5 | 4 | 1 | 2 | 1 | 5 | 3 | 1 | 22
  50,000 - <100,000 | 2 | 3 | 6 | 5 | 1 | 4 | 1 | 0 | 22
  >=100,000 | 2 | 11 | 2 | 7 | 3 | 12 | 14 | 11 | 62
HIV-1 log10 RNA [Mean (Standard Deviation); unit: log10 copies/mL] | 4.3 (0.5) | 4.9 (1.0) | 4.4 (0.8) | 4.9 (0.9) | 4.5 (1.4) | 4.5 (1.2) | 4.6 (1.1) | 4.6 (1.4) | 4.6 (1.1)
Class of Prior Antiretroviral Therapy (ART) [Count of Participants; unit: Participants] — Note: These categories are not mutually exclusive since some participants would have received multiple ARTs.
  Participants
    Nucleoside reverse transcriptase inhibitor (NRTI) | 23 | 23 | 14 | 17 | 6 | 30 | 29 | 23 | 165
    Non-nucleoside reverse transcriptase inhibitor (NNRTI) | 12 | 13 | 10 | 5 | 5 | 14 | 18 | 15 | 92
    Protease inhibitor (PI) | 18 | 17 | 10 | 15 | 5 | 25 | 28 | 20 | 138
    Fusion inhibitor (FI) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Grade 3 or Higher Adverse Events (AEs)
Description: All grade 3 or higher signs/symptoms, diagnoses, and laboratory AEs were included.
  AE grading was based on DAIDS AE Grading Table, Version 1.0, December 2004 (Clarification, August 2009).
  A 2-sided 95% Confidence Interval (CI) was calculated for the percentage using the binominal exact method.
Time Frame: From treatment initiation through Weeks 24 and 48
Population: Participants who received at least one dose of DTG and were deemed safety evaluable by the protocol team.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Cohort IIB: Children 6 to younger than 12 years of age who received DTG granules for suspension
  DTG granules for suspension initial starting dose at ~0.64 mg/kg with a maximum dose of 32 mg; orally once daily.
- Cohort IV: Children 6 months to younger than 2 years of age who received DTG granules for suspension
  DTG granules for suspension initial starting dose at ~0.64 mg/kg with a maximum dose of 32 mg; orally once daily.
Arm/Group | Cohort I | Cohort IIA | Cohort IIB | Cohort III | Cohort IV | Cohort III-DT | Cohort IV-DT | Cohort V-DT
Number analyzed (Participants) | 23 | 23 | 15 | 17 | 7 | 36 | 35 | 25
percentage of participants
  Through Week 24 | 4.3 [0.1 to 22.0] | 8.7 [1.1 to 28.0] | 6.7 [0.2 to 32.0] | 29.4 [10.3 to 56.0] | 57.1 [18.4 to 90.1] | 38.9 [23.1 to 56.5] | 42.9 [26.3 to 60.7] | 60 [38.7 to 78.9]
  Through Week 48 | 8.7 [1.1 to 28.0] | 17.4 [5.0 to 38.8] | 13.3 [1.7 to 40.5] | 35.3 [14.2 to 61.7] | 57.1 [18.4 to 90.1] | 41.7 [25.5 to 59.2] | 51.4 [34.0 to 68.6] | 64 [42.5 to 82.0]

2. Primary Outcome: Percentage of Participants With Grade 3 or Higher Adverse Events (AEs) Assessed as Related to Study Drug
Description: as for outcome 1
Time Frame: From treatment initiation through Weeks 24 and 48
Population: Participants who received at least one dose of DTG and were deemed safety evaluable by the protocol team.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort I | Cohort IIA | Cohort IIB | Cohort III | Cohort IV | Cohort III-DT | Cohort IV-DT | Cohort V-DT
Number analyzed (Participants) | 23 | 23 | 15 | 17 | 7 | 36 | 35 | 25
percentage of participants
  Through Week 24 | 0 [0.0 to 14.8] | 0 [0.0 to 14.8] | 0 [0.0 to 21.8] | 0 [0.0 to 19.5] | 14.3 [0.4 to 57.9] | 0 [0.0 to 9.7] | 0 [0.0 to 10.0] | 0 [0.0 to 13.7]
  Through Week 48 | 0 [0.0 to 14.8] | 0 [0.0 to 14.8] | 0 [0.0 to 21.8] | 0 [0.0 to 19.5] | 14.3 [0.4 to 57.9] | 0 [0.0 to 9.7] | 0 [0.0 to 10.0] | 0 [0.0 to 13.7]

3. Primary Outcome: Number of Participants With Permanent Discontinuation of Study Drug Due to Adverse Events (AEs) Assessed as Related to Study Drug
Description: Number of participants with permanent discontinuation of study drug due to AEs assessed by the site investigator as related to the study drug.
Time Frame: From treatment initiation through Weeks 24 and 48
Population: Participants who received at least one dose of DTG and were deemed safety evaluable by the protocol team.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort III: Children 2 to younger than 6 years of age who received DTG granules for suspension
  DTG granules for suspension initial starting dose at ~0.64 mg/kg with a maximum dose of 32 mg; orally once daily.
Arm/Group | Cohort I | Cohort IIA | Cohort IIB | Cohort III | Cohort IV | Cohort III-DT | Cohort IV-DT | Cohort V-DT
Number analyzed (Participants) | 23 | 23 | 15 | 17 | 7 | 36 | 35 | 25
Participants
  Through Week 24 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Through Week 48 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants Who Died
Description: Number of participants who died were summarized
Time Frame: From treatment initiation through Weeks 24 and 48
Population: Participants who received at least one dose of DTG and were deemed safety evaluable by the protocol team.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort I | Cohort IIA | Cohort IIB | Cohort III | Cohort IV | Cohort III-DT | Cohort IV-DT | Cohort V-DT
Number analyzed (Participants) | 23 | 23 | 15 | 17 | 7 | 36 | 35 | 25
Participants
  Through Week 24 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
  Through Week 48 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0

5. Primary Outcome: PK Parameter: Area-under-the-curve From 0 to 24 Hours (AUC0-24)
Description: Pharmacokinetic parameters were determined from plasma concentration-time profiles using non-compartmental methods (Phoenix WinNonlin 8.0 or current, Certara, Princeton, NJ). AUC0-24 was determined using linear up-log down estimation in WinNonlin.
Time Frame: One intensive PK visit between 5 and 10 days of DTG initiation. At intensive PK visit, blood samples were drawn pre-dose and at 1, 2, 3, 4, 6, 8 and 24 hours post dosing
Population: Participants with intensive pharmacokinetic (PK) data at the proposed dose for Cohorts I, IIA, III-DT, IV-DT, and V-DT.
Measure: Mean (Standard Deviation); unit: hr*mg/L
Groups:
- Cohort I: Adolescents 12 to younger than 18 years of age who received 50 mg DTG film-coated tablets orally once daily for those weighing ≥ 35kg.
- Cohort IIA: Children 6 to younger than 12 years of age who received 50 mg DTG film-coated tablets orally once daily for those weighing ≥ 35kg.
- Cohort III-DT: Children 2 to younger than 6 years of age who received weight band dosing at ~1 mg/kg of DTG dispersible tablet orally once daily.
- Cohort IV-DT: Children 6 months to younger than 2 years of age who received weight band dosing at ~1 mg/kg of DTG dispersible tablet orally once daily.
- Cohort V-DT: Infants 4 weeks to younger than 6 months of age who received weight band doing at ~1 mg/kg of DTG dispersible tablet orally once daily.
Arm/Group | Cohort I | Cohort IIA | Cohort III-DT | Cohort IV-DT | Cohort V-DT
Number analyzed (Participants) | 9 | 5 | 17 | 13 | 13
hr*mg/L | 52.98 (23.11) | 68.33 (43.33) | 63.16 (37.77) | 82.67 (47.05) | 71.45 (28.21)

6. Secondary Outcome: Percentage of Participants With Grade 3 or Higher Adverse Events (AEs)
Description: Percentage and exact 95% Confidence Interval (CI) of participants with Grade 3 or higher AEs. AEs were graded based on the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 1.0, December 2004, Clarification August 2009 (see References). All grade 3 or higher signs, symptoms, and laboratory toxicities were included.
Time Frame: From treatment initiation through Week 192. AEs after that time were censored.
Population: All participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort I | Cohort IIA | Cohort IIB | Cohort III | Cohort IV | Cohort III-DT | Cohort IV-DT | Cohort V-DT
Number analyzed (Participants) | 23 | 23 | 15 | 17 | 7 | 36 | 35 | 25
percentage of participants | 34.8 [16.4 to 57.3] | 30.4 [13.2 to 52.9] | 20 [4.3 to 48.1] | 52.9 [27.8 to 77.0] | 57.1 [18.4 to 90.1] | 58.3 [40.8 to 74.5] | 51.4 [34.0 to 68.6] | 64 [42.5 to 82.0]

7. Secondary Outcome: Percentage of Participants With Grade 3 or Higher Adverse Events (AEs) Assessed as Related to Study Drug
Description: Percentage and exact 95% Confidence Interval (CI) of participants with Grade 3 or higher AEs assessed by the site investigator as related to the study drug.
Time Frame: From treatment initiation through Week 192. AEs after that time were censored.
Population: All participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort I | Cohort IIA | Cohort IIB | Cohort III | Cohort IV | Cohort III-DT | Cohort IV-DT | Cohort V-DT
Number analyzed (Participants) | 23 | 23 | 15 | 17 | 7 | 36 | 35 | 25
percentage of participants | 0 [0.0 to 14.8] | 0 [0.0 to 14.8] | 0 [0.0 to 21.8] | 0 [0.0 to 19.5] | 14.3 [0.4 to 57.9] | 0 [0.0 to 9.7] | 0 [0.0 to 10.0] | 0 [0.0 to 13.7]

8. Secondary Outcome: Number of Participants With Permanent Discontinuation of Study Drug Due to Adverse Events (AEs) Assessed as Related to Study Drug
Description: as for outcome 3
Time Frame: From treatment initiation through Week 192. AEs after that time were censored.
Population: All participants
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort I | Cohort IIA | Cohort IIB | Cohort III | Cohort IV | Cohort III-DT | Cohort IV-DT | Cohort V-DT
Number analyzed (Participants) | 23 | 23 | 15 | 17 | 7 | 36 | 35 | 25
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Number of Participants Who Died
Description: Number of participants who died were summarized.
Time Frame: From treatment initiation through Week 192. AEs after that time were censored.
Population: All participants
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort I | Cohort IIA | Cohort IIB | Cohort III | Cohort IV | Cohort III-DT | Cohort IV-DT | Cohort V-DT
Number analyzed (Participants) | 23 | 23 | 15 | 17 | 7 | 36 | 35 | 25
Participants | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0

10. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA Less Than 400 Copies/ml
Description: Virologic responses were assessed at weeks 24 and 48 as percentages of participants and exact 95% Confidence Interval (CI). The virologic response or virologic failure was defined and calculated according to FDA's Snapshot algorithm.
Time Frame: Week 24 and Week 48
Population: Participants who received at least one dose of DTG.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort I | Cohort IIA | Cohort IIB | Cohort III | Cohort IV | Cohort III-DT | Cohort IV-DT | Cohort V-DT
Number analyzed (Participants) | 23 | 23 | 15 | 17 | 7 | 36 | 35 | 25
percentage of participants
  Week 24 | 82.6 [61.2 to 95] | 78.3 [56.3 to 92.5] | 100 [78.2 to 100] | 88.2 [63.6 to 98.5] | 71.4 [29 to 96.3] | 86.1 [70.5 to 95.3] | 88.6 [73.3 to 96.8] | 68 [46.5 to 85.1]
  Week 48 | 73.9 [51.6 to 89.8] | 78.3 [56.3 to 92.5] | 93.3 [68.1 to 99.8] | 94.1 [71.3 to 99.9] | 71.4 [29 to 96.3] | 86.1 [70.5 to 95.3] | 85.7 [69.7 to 95.2] | 72 [50.6 to 87.9]

11. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA Less Than 50 Copies/ml
Description: Virologic responses were assessed at weeks 24 and 48 as percentages of participants and exact 95% Confidence Interval (CI), The virologic response or virologic failure was defined and calculated according to FDA's Snapshot algorithm.
Time Frame: Week 24 and Week 48
Population: Participants who received at least one dose of DTG.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort I | Cohort IIA | Cohort IIB | Cohort III | Cohort IV | Cohort III-DT | Cohort IV-DT | Cohort V-DT
Number analyzed (Participants) | 23 | 23 | 15 | 17 | 7 | 36 | 35 | 25
percentage of participants
  Week 24 | 69.6 [47.1 to 86.8] | 60.9 [38.5 to 80.3] | 93.3 [68.1 to 99.8] | 58.8 [32.9 to 81.6] | 42.9 [9.9 to 81.6] | 61.1 [43.5 to 76.9] | 51.4 [34 to 68.6] | 32 [14.9 to 53.5]
  Week 48 | 60.9 [38.5 to 80.3] | 69.6 [47.1 to 86.8] | 93.3 [68.1 to 99.8] | 64.7 [38.3 to 85.8] | 42.9 [9.9 to 81.6] | 69.4 [51.9 to 83.7] | 65.7 [47.8 to 80.9] | 36 [18 to 57.5]

12. Secondary Outcome: PK Parameter: Plasma Concentration Observed at End of 24 Hour Dosing Interval (C24h)
Description: Determined from plasma concentration-time profiles using non-compartmental methods (Phoenix WinNonlin 8.0 or current, Certara, Princeton, NJ). C24h was taken directly from the observed concentration-time data or estimated using the elimination rate constant.
Time Frame: as for outcome 5
Population: Participants with intensive pharmacokinetic (PK) data at the proposed dose for Cohorts I, IIA, III-DT, IV-DT, and V-DT.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort I | Cohort IIA | Cohort III-DT | Cohort IV-DT | Cohort V-DT
Number analyzed (Participants) | 9 | 5 | 17 | 13 | 13
ng/mL | 1145.36 (659.65) | 1475.46 (1139.52) | 1065.12 (1112.46) | 1488.24 (1175.44) | 1765.19 (929.97)

13. Secondary Outcome: PK Parameter: Plasma Concentration Observed Immediately to Dosing of 24 Hour Dosing Interval (C0h)
Description: Determined from plasma concentration-time profiles using non-compartmental methods (Phoenix WinNonlin 8.0 or current, Certara, Princeton, NJ). C0h was taken directly from the observed concentration-time data.
Time Frame: as for outcome 5
Population: Participants with intensive pharmacokinetic (PK) data at the proposed dose for Cohorts I, IIA, III-DT, IV-DT, and V-DT.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort I | Cohort IIA | Cohort III-DT | Cohort IV-DT | Cohort V-DT
Number analyzed (Participants) | 9 | 5 | 17 | 13 | 13
ng/mL | 1429.09 (738.69) | 1508.44 (1271.93) | 944.22 (549.36) | 1584.29 (1388.27) | 1376.15 (1132.28)

14. Secondary Outcome: PK Parameter: Minimum Plasma Concentration (Cmin)
Description: Determined from plasma concentration-time profiles using non-compartmental methods (Phoenix WinNonlin 8.0 or current, Certara, Princeton, NJ) and were performed in real-time. Cmin was taken directly from the observed concentration-time data.
Time Frame: as for outcome 5
Population: Participants with intensive pharmacokinetic (PK) data at the proposed dose for Cohorts I, IIA, III-DT, IV-DT, and V-DT.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort I | Cohort IIA | Cohort III-DT | Cohort IV-DT | Cohort V-DT
Number analyzed (Participants) | 9 | 5 | 17 | 13 | 13
ng/mL | 1193.94 (668.76) | 1155.52 (1152.98) | 757.92 (439.83) | 1343.74 (1370.79) | 1213.68 (886.21)

15. Secondary Outcome: PK Parameter: Maximum Plasma Concentration (Cmax)
Description: Determined from plasma concentration-time profiles using non-compartmental methods (Phoenix WinNonlin 8.0 or current, Certara, Princeton, NJ). Cmax was taken directly from the observed concentration-time data.
Time Frame: as for outcome 5
Population: Participants with intensive pharmacokinetic (PK) data at the proposed dose for Cohorts I, IIA, III-DT, IV-DT, and V-DT.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort I | Cohort IIA | Cohort III-DT | Cohort IV-DT | Cohort V-DT
Number analyzed (Participants) | 9 | 5 | 17 | 13 | 13
ng/mL | 3945.97 (1499.34) | 5111.10 (2459.92) | 5530.16 (2466.62) | 6256.67 (2508.57) | 4832.58 (1679.69)

16. Secondary Outcome: PK Parameter: Apparent Clearance (CL/F)
Description: Determined from plasma concentration-time profiles using non-compartmental methods (Phoenix WinNonlin 8.0 or current, Certara, Princeton, NJ). CL/F was calculated as Dose/AUC.
Time Frame: as for outcome 5
Population: Participants with intensive pharmacokinetic (PK) data at the proposed dose for Cohorts I, IIA, III-DT, IV-DT, and V-DT.
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Cohort I | Cohort IIA | Cohort III-DT | Cohort IV-DT | Cohort V-DT
Number analyzed (Participants) | 9 | 5 | 17 | 13 | 13
L/h | 1.29 (1.03) | 1.11 (0.92) | 0.49 (0.31) | 0.23 (0.11) | 0.11 (0.05)

17. Secondary Outcome: PK Parameter: Apparent Volume of Distribution (Vz/F)
Description: Determined from plasma concentration-time profiles using non-compartmental methods (Phoenix WinNonlin 8.0 or current, Certara, Princeton, NJ). Vz/F was calculated as Dose/(ke x AUC).
Time Frame: as for outcome 5
Population: Participants with intensive pharmacokinetic (PK) data at the proposed dose for Cohorts I, IIA, III-DT, IV-DT, and V-DT.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Cohort I | Cohort IIA | Cohort III-DT | Cohort IV-DT | Cohort V-DT
Number analyzed (Participants) | 9 | 5 | 17 | 13 | 13
L | 21.95 (13.71) | 19.11 (16.51) | 5.75 (3.66) | 3.19 (1.50) | 2.37 (1.04)

18. Secondary Outcome: PK Parameter: Terminal Half-life (t1/2)
Description: Determined from plasma concentration-time profiles using non-compartmental methods (Phoenix WinNonlin 8.0 or current, Certara, Princeton, NJ). t1/2 was calculated as ln(2)/ke.
Time Frame: as for outcome 5
Population: Participants with intensive pharmacokinetic (PK) data at the proposed dose for Cohorts I, IIA, III-DT, IV-DT, and V-DT.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Cohort I | Cohort IIA | Cohort III-DT | Cohort IV-DT | Cohort V-DT
Number analyzed (Participants) | 9 | 5 | 17 | 13 | 13
h | 13.21 (5.51) | 12.22 (2.63) | 9.10 (3.40) | 9.93 (2.58) | 16.85 (8.22)

19. Secondary Outcome: Summary of Changes in CD4 Count From Baseline
Description: The median differences between CD4 count at Week 24 and 48 minus at the Day 0 (baseline), and Interquartile Ranges (IQRs) are presented.
Time Frame: Measured at Day 0, Week 24, and Week 48
Population: Participants who received at least one dose of DTG. Study participants who had non-missing values were summarized.
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Groups:
- Cohort V-DT: Infants 4 weeks to younger than 6 months of age who received DTG dispersible tablets.
  DTG dispersible tablets initial starting dose of ~0.8 mg/kg with a maximum dose of 30 mg; orally once daily.
Arm/Group | Cohort I | Cohort IIA | Cohort IIB | Cohort III | Cohort IV | Cohort III-DT | Cohort IV-DT | Cohort V-DT
Number analyzed (Participants) | 23 | 23 | 15 | 17 | 7 | 36 | 35 | 25
cells/mm^3
  From baseline to Week 24: number analyzed (Participants) | 23 | 21 | 15 | 17 | 6 | 33 | 33 | 23
  From baseline to Week 24 | 63 [-56 to 180] | 209 [30 to 403] | 268 [142 to 372] | 199 [-59 to 644] | 472 [-20 to 883] | 249 [47 to 535] | 110 [-284 to 434] | 441 [-114 to 1023]
  From baseline to Week 48: number analyzed (Participants) | 22 | 21 | 15 | 16 | 5 | 33 | 33 | 22
  From baseline to Week 48 | 84 [-81 to 238] | 387 [49 to 575] | 246 [160 to 466] | 134.5 [-183.5 to 569.5] | 577 [135 to 777] | 191 [-202 to 541] | -1 [-449 to 577] | 721 [-114 to 972]

20. Secondary Outcome: Summary of Changes in CD4 Percent From Baseline
Description: The median differences between CD4 percent at Week 24 and 48 minus at the Day 0 (baseline), and Interquartile Ranges (IQRs) are presented.
Time Frame: Measured at Day 0, Week 24, and Week 48
Population: Participants who received at least one dose of DTG. Study participants who had non-missing values were summarized.
Measure: Median (Inter-Quartile Range); unit: Percentage of total lymphocytes
Arm/Group | Cohort I | Cohort IIA | Cohort IIB | Cohort III | Cohort IV | Cohort III-DT | Cohort IV-DT | Cohort V-DT
Number analyzed (Participants) | 23 | 23 | 15 | 17 | 7 | 36 | 35 | 25
Percentage of total lymphocytes
  From baseline to Week 24: number analyzed (Participants) | 23 | 21 | 15 | 17 | 6 | 33 | 33 | 23
  From baseline to Week 24 | 4.9 [1 to 8] | 8 [5 to 11] | 6 [3.3 to 9.1] | 6 [4.5 to 9] | 5.7 [3.9 to 8.1] | 6.1 [3.4 to 10.9] | 6 [2.5 to 12] | 5.1 [1 to 10]
  From baseline to Week 48: number analyzed (Participants) | 22 | 21 | 15 | 16 | 5 | 33 | 33 | 22
  From baseline to Week 48 | 4.7 [0 to 9.4] | 9 [7 to 14] | 9.2 [5 to 11.9] | 5.6 [1.5 to 11] | 9.9 [8.5 to 10] | 9.1 [4.4 to 13.4] | 8.8 [0.7 to 14] | 9.7 [4.1 to 11]

21. Secondary Outcome: Summary of Changes in CD8 Count From Baseline
Description: The median differences between CD8 count at Week 24 and 48 minus at the Day 0 (baseline), and Interquartile Ranges (IQRs) are presented.
Time Frame: Measured at Day 0, Week 24, and Week 48
Population: Participants who received at least one dose of DTG. Study participants who had non-missing values were summarized.
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | Cohort I | Cohort IIA | Cohort IIB | Cohort III | Cohort IV | Cohort III-DT | Cohort IV-DT | Cohort V-DT
Number analyzed (Participants) | 23 | 23 | 15 | 17 | 7 | 36 | 35 | 25
cells/mm^3
  From baseline to Week 24: number analyzed (Participants) | 23 | 21 | 15 | 17 | 6 | 33 | 33 | 23
  From baseline to Week 24 | -36 [-371 to 30] | -147 [-804 to 30] | -43 [-247 to 151] | -282 [-533 to 176] | 223 [-592 to 668] | -395 [-732 to 69] | -813 [-2013 to -65] | -210 [-1206 to 910]
  From baseline to Week 48: number analyzed (Participants) | 22 | 21 | 15 | 16 | 5 | 33 | 33 | 22
  From baseline to Week 48 | -52.5 [-365 to 105] | -117 [-607 to 131] | -126 [-302 to 166] | -431.5 [-782 to -169.5] | -376 [-411 to 21] | -464 [-1013 to -94] | -1242 [-2433 to -280] | -442 [-1435 to 870]

22. Secondary Outcome: Summary of Changes in CD8 Percent From Baseline
Description: The median differences between CD8 percent at Week 24 and 48 minus at the Day 0 (baseline), and Interquartile Ranges (IQRs) are presented.
Time Frame: Measured at Day 0, Week 24, and Week 48
Population: Participants who received at least one dose of DTG. Study participants who had non-missing values were summarized.
Measure: Median (Inter-Quartile Range); unit: Percentage of total lymphocytes
Arm/Group | Cohort I | Cohort IIA | Cohort IIB | Cohort III | Cohort IV | Cohort III-DT | Cohort IV-DT | Cohort V-DT
Number analyzed (Participants) | 23 | 23 | 15 | 17 | 7 | 36 | 35 | 25
Percentage of total lymphocytes
  From baseline to Week 24: number analyzed (Participants) | 23 | 21 | 15 | 17 | 6 | 33 | 33 | 23
  From baseline to Week 24 | -5 [-9.7 to -2.3] | -10 [-17.4 to -6] | -7 [-9.2 to -4] | -6.8 [-9.9 to 2.5] | -2 [-4.1 to 3.5] | -3 [-9 to 0.1] | -4.2 [-9.9 to -1.3] | -4 [-10.2 to 2]
  From baseline to Week 48: number analyzed (Participants) | 22 | 21 | 15 | 16 | 5 | 33 | 33 | 22
  From baseline to Week 48 | -6 [-12 to -2.4] | -11.4 [-22 to -7] | -8 [-15 to -5] | -6.5 [-14.5 to -3] | -1.8 [-4 to 0.3] | -6.5 [-10 to -1.9] | -9 [-15.2 to -4.9] | -3.5 [-11.5 to 1.7]

23. Secondary Outcome: Genotypic Measures of Resistance to Integrase
Description: Genes were sequenced and compared to a reference sequence to identify mutations
Time Frame: At baseline
Population: All participants with a confirmed decrease in HIV RNA of < 1.0 log10 at or after week 12 unless the HIV RNA is < 400 copies/mL, or a confirmed HIV RNA > 400 copies/mL starting at Week 24 or beyond on 2 consecutive measurements at least 1 week and within 4 weeks apart
Measure: Count of Participants; unit: Participants
Groups:
- All VF Participants: All participants with virological failure
Arm/Group | All VF Participants
Number analyzed (Participants) | 56
Participants
  A128T | 2
  Gene not found | 3
  L74I | 7
  L74I,S230N | 1
  S230N | 1
  T97A | 1
  V151I | 1
  None | 40

24. Secondary Outcome: Genotypic Measures of Resistance to Integrase
Description: Genes were sequenced and compared to a reference sequence to identify mutations
Time Frame: at virological failure visit at or prior to Week 192
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | All VF Participants
Number analyzed (Participants) | 56
Participants
  A128T | 1
  A128T,S153AFSV | 1
  E138AEKT,E138T,S147G,S147GS,R263K,R263KR | 1
  E138K,Q148K | 1
  E157Q | 1
  E92EG,T97A,N155H,N155HN | 1
  E92EQ,G118GR | 1
  H51HY | 1
  L74I | 4
  L74I,G118R | 1
  L74I,S230N | 1
  L74M,G118R | 1
  R263K | 1
  S230N | 1
  T66I,G118R,E138A | 1
  T66I,L74I,G118R | 1
  T97A,G118R,E138EK,S147G,V151I,N155H | 1
  missing | 11
  None | 25

25. Secondary Outcome: Genotypic Measures of Resistance to Protease
Description: Genes were sequenced and compared to a reference sequence to identify mutations
Time Frame: at baseline
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | All VF Participants
Number analyzed (Participants) | 56
Participants
  A71T | 1
  D30N,A71T,N88D | 1
  D30N,M46I,Q58EQ,A71T,N88D | 1
  I84V | 1
  K20I | 2
  K20I,V82I | 1
  K20R | 8
  K20R,A71T | 1
  K20R,L33F,M46I,I50V,I54V,T74P,V82A | 1
  K20R,T74S | 1
  K20R,T74S,V82A | 1
  K20T,V82I | 1
  K43T,A71T,V82A | 1
  L10I,K20KR,M46LM,I54IL,A71AV,V82AFSV | 3
  L10I | 1
  L10V | 2
  T74S | 3
  None | 26

26. Secondary Outcome: Genotypic Measures of Resistance to Protease
Description: Genes were sequenced and compared to a reference sequence to identify mutations
Time Frame: at virological failures at or prior to Week 192
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | All VF Participants
Number analyzed (Participants) | 56
Participants
  A71T | 2
  D30N,A71T,N88D | 1
  D30N,M46I,Q58E,Q58EQ,A71T,N88D | 1
  I84V | 1
  K20I | 1
  K20R | 7
  K20R,T74S | 1
  K20R,T74S,V82A | 1
  K20T,V82I | 1
  L10I | 6
  L10I,K20R | 1
  L10I,K43T,I54V,A71T,V82A | 1
  L10I,L10IV | 1
  L10IL,K20KR,L33FL,M46IM,I50IV,I54IV,T74PT,V82AV | 1
  L10V | 2
  L10V,K20IV,K20V | 1
  T74S | 3
  V11IV,K20I,V82I | 1
  missing | 8
  None | 15

27. Secondary Outcome: Genotypic Measures of Resistance to Reverse Transcriptase
Description: Genes were sequenced and compared to a reference sequence to identify mutations
Time Frame: at baseline
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | All VF Participants
Number analyzed (Participants) | 56
Participants
  A62V,K65R,S68G,K70R,V75I,F77L,K101Q,K103N,F116Y,Q151M,P225H | 1
  D67DN,K238R | 1
  D67DN,V179I,V179IV,M184V,K219Q,N348I | 1
  E138A | 1
  E44D,K103N,M184V | 1
  K103N | 4
  K103N,M184V | 1
  K103N,M184V,M184MV | 1
  K103N,P225H | 1
  K103N,V179I | 1
  K103N,V179I,M184V | 1
  K103N,Y181C | 1
  K103S,V179I,G190A,Y318F | 1
  K65R,V106M,G190A | 1
  K70KR,T215F,T215FIST,K238R | 1
  L74LV,Y181CY,M184V | 1
  L74V,K103N,E138G,M184V,M230L | 1
  L74V,V106M,Y181C | 1
  M184V | 2
  M184V,H221Y | 1
  M184V,K238R | 1
  M41L,D67N,T69N,K70R,L74I,A98G,M184V,T215F,K219Q,K238R | 1
  M41L,K101E,V179I,M184V,G190A,T215F | 1
  M41L,T215L | 1
  S68G,K103N,E138Q,M184V,Y318F | 1
  S68G,V106I,K238R | 1
  S68G,V90I,K103N,V179I | 1
  T69D | 1
  V118I,E138A | 1
  V118IV,V179I,M184V | 1
  V179E,P225H | 1
  V179I | 1
  V179I,M184V | 2
  V179I,M184V,G190A,K219R | 1
  V179I,M184V,K238R | 1
  V179I,M184V,Y188L | 1
  V179S | 1
  V75M,K103N | 1
  V90I | 2
  Y181C | 1
  None | 10

28. Secondary Outcome: Genotypic Measures of Resistance to Reverse Transcriptase
Description: Genes were sequenced and compared to a reference sequence to identify mutations
Time Frame: at virologic failure at or prior to Week 192
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | All VF Participants
Number analyzed (Participants) | 56
Participants
  101i,V179I,M184V | 1
  A62V,K65R,S68G,K70R,V75I,F77L,K101Q,K103N,F116Y,Q151M,P225H | 1
  D67N,K219Q,N348I | 1
  E138A | 1
  E44D,E44DE,K103N,M184V | 1
  E44DE | 1
  K103KN,K103N,M184V | 1
  K103N | 4
  K103N,M184V | 1
  K103N,V179I | 1
  K103N,V179I,M184V | 1
  K103S,M184V,G190A,Y318F | 1
  K238R | 2
  K238R,M41LM,D67DN,T69NT,K70KR,L74IL,A98AG,M184MV,T215FIST,K219Q,M230IM | 1
  L74IL,L74V,K103N,E138G,M184V,M230L | 1
  M184V | 3
  M184V,H221Y | 1
  M184V,K238R | 1
  M41L,T215FL | 1
  M41LM,M184V,S68G,S68GS,Y181CY,M184MV | 1
  S68G,V106I,K238R | 1
  S68G,V90I,K103N,V179I,M184V | 1
  S68GS,K103KN,K238KR,K238R | 1
  T69NT,K103N,P225H | 1
  V106M,Y181C,P236LP | 1
  V179D,V179DV,G190A,G190AG | 1
  V179E,P225H | 1
  V179I | 1
  V179I,M184V | 1
  V179I,M184V,G190A,K219R | 1
  V179I,M184V,K238R | 1
  V179I,M184V,Y188L | 1
  V179S,M184V | 1
  V75M,K103N | 1
  V90I | 1
  missing | 6
  None | 9

29. Secondary Outcome: Phenotypic Measures of Resistance
Description: The participant viral culture is considered to be reduced susceptibility if more DTG is needed to inactivate 50% of the participant viral culture compared to the control viral specimen
Time Frame: Whenever virological failures took place from baseline to week 192
Population: Protocol defined virological failure population for which drug susceptibility was measured
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort I | Cohort IIA | Cohort IIB | Cohort III | Cohort IV | Cohort III-DT | Cohort IV-DT | Cohort V-DT
Number analyzed (Participants) | 11 | 5 | 1 | 3 | 3 | 10 | 11 | 12
Participants
  Sensitive to DTG | 8 | 4 | 0 | 2 | 0 | 5 | 4 | 9
  Reduced susceptibility to DTG | 2 | 0 | 1 | 0 | 1 | 1 | 0 | 0
  missing | 1 | 1 | 0 | 1 | 2 | 4 | 7 | 3

30. Secondary Outcome: Worst Case CDC HIV Classification Status
Description: Disease progression as measured by change from baseline to the worst case CDC HIV classification status
Time Frame: From baseline through Week 192
Population: All participants enrolled into the study
Measure: Count of Participants; unit: Participants
Groups:
- Not Symptomatic: The worst-case CDC HIV classification status was not symptomatic (<13 years of age)
- Mildly Symptomatic: The worst-case CDC HIV classification status is mildly symptomatic (<13 years of age)
- Moderately Symptomatic: The worst-case CDC HIV classification status was moderately symptomatic (<13 years of age)
- Severely Symptomatic: The worst-case CDC HIV classification status was severely symptomatic (<13 years of age)
- Stage III: The worst-case CDC HIV classification status was Stage III (>= 13 years of age)
- Stage I or II: The worst-case CDC HIV classification status was Stage I (acute HIV infection) or II (chronic HIV infection) (>= 13 years of age)
Arm/Group | Not Symptomatic | Mildly Symptomatic | Moderately Symptomatic | Severely Symptomatic | Stage III | Stage I or II
Number analyzed (Participants) | 74 | 37 | 21 | 32 | 7 | 10
Participants
  Not symptomatic at entry | 74 | 0 | 1 | 0 | 0 | 0
  Mildly symptomatic at entry | 0 | 37 | 0 | 0 | 0 | 0
  Moderately symptomatic at entry | 0 | 0 | 20 | 1 | 0 | 0
  Severely symptomatic at entry | 0 | 0 | 0 | 31 | 0 | 0
  Stage III at entry | 0 | 0 | 0 | 0 | 7 | 0
  Stage I or II at entry | 0 | 0 | 0 | 0 | 0 | 10

ADVERSE EVENTS:
Time Frame: From study entry to completion of follow-up by Week 192 or longer, for participants on long-term follow-up. Five, 4, 3, 1 and 1 participants completed visit week 216, 228, 240, 278 and 284, respectively; all follow-up was included.
Description: AEs were summarized for participants who received at least one dose of Dolutegravir (DTG). AE severity grading was based on the DAIDS AE Grading Table, Version 1.0. SAEs were reported according to DAIDS EAE Manual V2.0.
Groups:
- Cohort III-DT: Children 2 to younger than 6 years of age who received DTG dispersible tablets. DTG dispersible tables initial starting dose of ~0.8 mg/kg with a maximum dose of 30 mg; orally once daily.
- Cohort IV-DT: Children 6 months to younger than 2 years of age who received DTG dispersible tablets.
  DTG dispersible tables initial starting dose of ~1.25 mg/kg with a maximum dose of 30 mg; orally once daily.
- Cohort V-DT: Infants 4 weeks to younger than 6 months of age who received DTG dispersible tablets.
  DTG dispersible tables initial starting dose of ~1.25 mg/kg with a maximum dose of 30 mg; orally once daily.
Arm/Group | Cohort I | Cohort IIA | Cohort IIB | Cohort III | Cohort IV | Cohort III-DT | Cohort IV-DT | Cohort V-DT
All-Cause Mortality (participants affected / at risk) | 0/23 | 1/23 | 0/15 | 0/17 | 0/7 | 1/36 | 1/35 | 0/25
Serious Adverse Events (participants affected / at risk) | 8/23 | 5/23 | 1/15 | 8/17 | 2/7 | 12/36 | 8/35 | 2/25
Other Adverse Events (participants affected / at risk) | 23/23 | 23/23 | 15/15 | 17/17 | 7/7 | 36/36 | 35/35 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort I (N=23) | Cohort IIA (N=23) | Cohort IIB (N=15) | Cohort III (N=17) | Cohort IV (N=7) | Cohort III-DT (N=36) | Cohort IV-DT (N=35) | Cohort V-DT (N=25)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Drowning (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Atypical mycobacterial lymphadenitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bacterial sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Disseminated mycobacterium avium complex infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
Gastroenteritis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ophthalmic herpes simplex (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pelvic inflammatory disease (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Plasmodium falciparum infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1
Pneumonia adenoviral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinusitis bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinea versicolour (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Viral rash (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood glucose decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retinoblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Febrile convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abnormal behaviour (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acquired hydrocele (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abortion induced (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort I (N=23) | Cohort IIA (N=23) | Cohort IIB (N=15) | Cohort III (N=17) | Cohort IV (N=7) | Cohort III-DT (N=36) | Cohort IV-DT (N=35) | Cohort V-DT (N=25)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 1 | 2 | 2 | 3
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 7 | 7 | 3 | 2 | 2 | 6 | 1 | 2
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Craniosynostosis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Phimosis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 2 | 4 | 2 | 4 | 1 | 5 | 0 | 0
Noninfective myringitis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Otorrhoea (Ear and labyrinth disorders) | 0 | 3 | 1 | 2 | 0 | 2 | 2 | 1
Tympanic membrane disorder (Ear and labyrinth disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Tympanic membrane hyperaemia (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chalazion (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Conjunctival hyperaemia (Eye disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Conjunctival pallor (Eye disorders) | 2 | 1 | 0 | 1 | 2 | 1 | 2 | 3
Eye discharge (Eye disorders) | 1 | 0 | 1 | 3 | 1 | 0 | 5 | 1
Eye movement disorder (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye opacity (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1
Ocular hyperaemia (Eye disorders) | 1 | 1 | 2 | 0 | 1 | 2 | 4 | 1
Pterygium (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Scleritis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 7 | 1 | 2 | 2 | 1 | 7 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 4 | 3 | 1 | 1 | 0 | 0 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Anal erythema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Anal pruritus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 1
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 1 | 2 | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 8 | 6 | 2 | 9 | 4 | 10 | 19 | 6
Dysphagia (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Gingival ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infantile vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Lip pain (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Lip ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 8 | 1 | 2 | 1 | 0 | 1 | 0 | 0
Noninfective gingivitis (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral disorder (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 0
Oral mucosal eruption (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral mucosal erythema (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1
Toothache (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 6 | 4 | 6 | 7 | 3 | 11 | 14 | 8
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Fatigue (General disorders) | 3 | 2 | 1 | 0 | 0 | 1 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 1 | 0 | 0 | 3 | 4 | 0
Influenza like illness (General disorders) | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Medical device site pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 3 | 2 | 1 | 2 | 0 | 2 | 1 | 0
Pyrexia (General disorders) | 8 | 7 | 5 | 9 | 6 | 18 | 13 | 7
Ulcer (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 1 | 0 | 2 | 1 | 2 | 0 | 1
Allergy to arthropod bite (Immune system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Immune reconstitution inflammatory syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Acarodermatitis (Infections and infestations) | 2 | 0 | 2 | 2 | 1 | 2 | 4 | 1
Adenoiditis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Ascariasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bacterial vaginosis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Balanitis candida (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Body tinea (Infections and infestations) | 1 | 0 | 2 | 1 | 1 | 5 | 3 | 2
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 2 | 2 | 1 | 0 | 1 | 0 | 0
Bronchitis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 1 | 1 | 1 | 1 | 5 | 0
Enterobiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 1 | 5 | 1 | 3 | 8 | 2
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Giardiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
HIV-associated neurocognitive disorder (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Helminthic infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Herpangina (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Impetigo (Infections and infestations) | 1 | 3 | 1 | 4 | 3 | 6 | 4 | 1
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lice infestation (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0
Measles (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Molluscum contagiosum (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0 | 2 | 3 | 3 | 1 | 0
Oral candidiasis (Infections and infestations) | 2 | 0 | 1 | 0 | 1 | 2 | 4 | 2
Oral herpes (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 2 | 2 | 0 | 4 | 0 | 5 | 4 | 2
Otitis media chronic (Infections and infestations) | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0
Parasitic gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0
Pharyngitis (Infections and infestations) | 3 | 2 | 3 | 4 | 0 | 8 | 5 | 2
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 3 | 1 | 1 | 0 | 1 | 0 | 2
Pustule (Infections and infestations) | 2 | 2 | 1 | 1 | 1 | 1 | 0 | 2
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 5 | 2
Schistosomiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Septic rash (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Sinusitis bacterial (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 2 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tinea capitis (Infections and infestations) | 0 | 4 | 0 | 0 | 1 | 5 | 5 | 2
Tinea faciei (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 4 | 1 | 0
Tinea infection (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Tinea versicolour (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 2 | 3 | 0 | 5 | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 2 | 9 | 10 | 4
Upper respiratory tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 2 | 0 | 2 | 5 | 1
Varicella (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 1
Viral infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Adverse event following immunisation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Scar (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 2 | 2 | 0 | 0 | 1 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Skin wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 5 | 8 | 4 | 5 | 3 | 7 | 2 | 4
Aspartate aminotransferase increased (Investigations) | 5 | 7 | 3 | 8 | 3 | 12 | 8 | 3
Blood albumin decreased (Investigations) | 3 | 4 | 2 | 2 | 2 | 6 | 12 | 11
Blood alkaline phosphatase increased (Investigations) | 2 | 5 | 4 | 3 | 3 | 11 | 7 | 6
Blood bicarbonate decreased (Investigations) | 11 | 10 | 6 | 13 | 6 | 33 | 34 | 23
Blood bilirubin increased (Investigations) | 5 | 6 | 3 | 1 | 0 | 1 | 0 | 0
Blood calcium decreased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Blood calcium increased (Investigations) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Blood cholesterol increased (Investigations) | 2 | 2 | 1 | 1 | 1 | 6 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 2
Blood glucose decreased (Investigations) | 8 | 12 | 7 | 8 | 3 | 10 | 10 | 5
Blood glucose increased (Investigations) | 2 | 4 | 2 | 1 | 3 | 13 | 13 | 6
Blood phosphorus decreased (Investigations) | 3 | 2 | 2 | 0 | 1 | 3 | 5 | 5
Blood potassium decreased (Investigations) | 4 | 2 | 1 | 2 | 1 | 2 | 4 | 0
Blood potassium increased (Investigations) | 0 | 1 | 1 | 3 | 1 | 10 | 11 | 14
Blood pressure diastolic increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 3 | 0 | 0
Blood pressure increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood pressure systolic increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0
Blood sodium decreased (Investigations) | 6 | 8 | 9 | 8 | 7 | 24 | 27 | 14
Blood sodium increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 3 | 0 | 4
Blood urine present (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Breath sounds abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1
Cardiac murmur (Investigations) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 6 | 0 | 5 | 3 | 14 | 24 | 20
Lipase increased (Investigations) | 2 | 2 | 2 | 3 | 2 | 6 | 8 | 3
Low density lipoprotein increased (Investigations) | 1 | 2 | 1 | 0 | 0 | 5 | 0 | 0
Neutrophil count decreased (Investigations) | 4 | 6 | 7 | 6 | 3 | 19 | 20 | 19
Platelet count decreased (Investigations) | 2 | 0 | 2 | 3 | 0 | 2 | 1 | 2
Urine output decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 2 | 0 | 3 | 0 | 2 | 3 | 0
White blood cell count decreased (Investigations) | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 7 | 3 | 3 | 5 | 5 | 4 | 10 | 4
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0
Feeding disorder (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2
Poor feeding infant (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0
Underweight (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 3 | 0 | 1 | 0 | 1 | 0 | 0
Weight gain poor (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 2 | 1 | 0 | 0 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 1 | 1 | 1 | 0 | 3 | 2 | 0
Clonus (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 4 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 8 | 6 | 5 | 3 | 0 | 4 | 1 | 0
Hypertonia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Meningism (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Motor developmental delay (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle spasticity (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Adjustment disorder with disturbance of conduct (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Attention deficit hyperactivity disorder (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Reading disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 2 | 2 | 0 | 2 | 0 | 0 | 2 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 2 | 0 | 2 | 0 | 1 | 0 | 1
Proteinuria (Renal and urinary disorders) | 2 | 0 | 0 | 2 | 0 | 1 | 1 | 1
Genital rash (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Intermenstrual bleeding (Reproductive system and breast disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Perineal erythema (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Bronchial wall thickening (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0
Childhood asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 15 | 8 | 15 | 6 | 29 | 21 | 15
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 2 | 2 | 2 | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mouth breathing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 10 | 10 | 5 | 6 | 4 | 8 | 5 | 5
Nasal discharge discolouration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 11 | 5 | 4 | 2 | 0 | 10 | 2 | 0
Oropharyngeal plaque (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 1 | 1 | 1 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 3 | 2 | 6 | 8 | 3
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 2 | 2 | 3 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 2 | 4 | 1 | 10 | 1 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 7 | 8 | 8 | 10 | 5 | 15 | 11 | 6
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 3 | 3 | 4 | 2 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 3
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2 | 0 | 2 | 1 | 0
Tonsillar inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 1 | 2 | 1 | 0
Use of accessory respiratory muscles (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0 | 3 | 1 | 3 | 4 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 0 | 2 | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0 | 0 | 1 | 2 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 4 | 1 | 0 | 0 | 1 | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 1 | 0 | 1 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 1 | 0 | 0 | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 2 | 0 | 3 | 0 | 1
Macule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 2 | 2 | 2 | 5 | 2 | 3 | 4 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 6 | 3 | 0 | 1 | 6 | 7 | 0
Rash (Skin and subcutaneous tissue disorders) | 5 | 7 | 6 | 3 | 2 | 11 | 13 | 7
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 4 | 4 | 1
Scab (Skin and subcutaneous tissue disorders) | 0 | 3 | 1 | 1 | 0 | 2 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 3 | 2 | 0 | 0 | 0 | 0 | 0
Skin plaque (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pallor (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights

DOCUMENTS (5):
  • Study Protocol: Protocol V5.0 (2018-07-12): https://cdn.clinicaltrials.gov/large-docs/47/NCT01302847/Prot_001.pdf
  • Study Protocol: Protocol V5.0_Letter of Amendment 1 (2020-06-10): https://cdn.clinicaltrials.gov/large-docs/47/NCT01302847/Prot_002.pdf
  • Statistical Analysis Plan: Primary Statistical Analysis Plan (2021-04-22): https://cdn.clinicaltrials.gov/large-docs/47/NCT01302847/SAP_003.pdf
  • Statistical Analysis Plan: Pharmacokinetics (PK) Statistical Analysis Plan (2019-04-08): https://cdn.clinicaltrials.gov/large-docs/47/NCT01302847/SAP_004.pdf
  • Informed Consent Form (2018-07-12): https://cdn.clinicaltrials.gov/large-docs/47/NCT01302847/ICF_000.pdf